CLINICAL TRIAL: NCT07369414
Title: Environmental Reservoirs of Non-tuberculous Mycobacteria in Cystic Fibrosis Households: A Case-control Study of Exposure Risk at Home
Acronym: NTMecoCF
Status: Recruiting | Type: Observational
Sponsor: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Alexander Mischnik, Prof. Dr. med. Alexander Mischnik, Research Center Borstel
Other Study IDs: NTMecoCF
Record Dates: First submitted 2026-01-16; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis (CF); Mucoviscidosis; Non-Tuberculous Mycobacteria; Mycobacterium Abscessus Infection
Keywords: Environmental reservoirs; Household water systems; Microbial exposure; Whole-genome sequencing; Environmental risk factors
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous | interventions — Whole Genome Sequencing; Culture Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mycobacterial strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: 60 CF patients with a confirmed current or previously diagnosed NTM infection (according to ATS/IDSA criteria)
  Interventions: Other: Multi-modal NTM diagnostic including PCR, WGS, culture
- Control group: 60 CF patients without a known or previously diagnosed NTM infection (according to ATS/IDSA criteria)
  Interventions: Other: Multi-modal NTM diagnostic including PCR, WGS, culture

INTERVENTIONS:
Other: Multi-modal NTM diagnostic including PCR, WGS, culture — Environmental samples from participants' households (e.g., water, dust, and soil) will be collected and tested for the presence of NTM. Analyses will be performed using PCR, culture-based methods, whole-genome sequencing (WGS), and subsequent bioinformatic analyses. In addition, available clinical NTM isolates from previous or future routine diagnostics will be included. If genomic sequencing has not yet been performed for these isolates, retrospective molecular genetic analysis (e.g., by WGS) will be conducted within the study to enable comparison with environmental isolates.

SUMMARY:
This multicenter, non-interventional case-control study investigates whether household environmental reservoirs, particularly water systems, are associated with non-tuberculous mycobacterial (NTM) infections in people with cystic fibrosis. Environmental samples from the homes of CF patients with and without NTM infection will be analyzed and genetically compared with available clinical isolates, alongside assessment of environmental risk factors, to improve understanding of exposure pathways and inform future prevention strategies.

DETAILED DESCRIPTION:
This multicenter, non-interventional case-control study investigates whether domestic environmental reservoirs-particularly household water systems-contribute to non-tuberculous mycobacterial (NTM) infections in people with cystic fibrosis (CF). Approximately 120 CF patients from several centers in Germany will be enrolled, including 60 patients with a current or previous pulmonary NTM infection and 60 CF patients without known NTM infection as controls.

Environmental samples (water, dust, and soil) will be collected from participants' households and analyzed for the presence of NTM using culture-based methods, PCR, and whole-genome sequencing. These findings will be compared between case and control households, and genetic similarity between environmental NTM isolates and available clinical isolates from the same patients will be assessed. In addition, standardized questionnaires will capture environmental and behavioral risk factors associated with NTM occurrence.

The study is purely observational and relies on clinical data and isolates obtained through routine CF care, with no additional medical procedures for participants. Over a follow-up period of up to three years, newly occurring NTM infections in initially unaffected patients will be documented. The results aim to improve understanding of environmental exposure risks for NTM in CF and to provide evidence for future prevention strategies and potential guideline recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis (CF)
* No age restriction (including minors with consent from legal guardians)
* Written informed consent to participate in the study (or consent provided by a legal guardian for minors)
* In the case of an NTM infection: diagnosis according to ATS/IDSA criteria and availability of a clinical NTM isolate

Exclusion Criteria:

* Lack of capacity to provide informed consent, refusal to participate, or withdrawal of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises 120 individuals with a confirmed diagnosis of cystic fibrosis recruited from multiple centers in Germany. Participants include both adults and minors (with consent from legal guardians) and are divided equally into a case group of patients with a current or prior pulmonary NTM infection and a control group of patients without a known history of NTM infection. All participants provide written informed consent, and clinical data and isolates are obtained exclusively from routine care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NTM in environmental samples | 2030
  Proportion of households of CF patients with and without NTM infection in which at least one (clinically relevant) NTM is detected in environmental samples (water, dust, soil).
Difference in NTM prevalence between case and control groups | 2030
  Statistically significant difference in the frequency of NTM detection (clinically relevant and/or all NTM) in environmental samples between case group and control group.
Genetic concordance between environmental and patient isolates | 2030
  Evidence of genetic relatedness (e.g., cgMLST clustering) between NTM detected in the household environment and clinical isolates from the same individual.

SECONDARY OUTCOMES:
Characterization of NTM species from environmental samples | 2030
  Identification and taxonomic classification of NTM isolates using WGS, including typing (e.g., subspecies assignment for M. avium).
Identification of environmental and behavioral factors associated with NTM detection | 2030
  Determination of significant risk factors (e.g., use of specific water sources, pet ownership, hygiene practices) based on questionnaire data and multivariable analyses.
Long-term outcomes (control group only) | 2030
  Proportion of patients without an initial NTM infection who develop a clinically relevant NTM infection during the follow-up period (up to 30 months), potentially in association with prior detection of NTM in the household environment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mischnik, Prof. Dr. med., Principal Investigator — National and WHO-Supranational Reference Center for Mycobacteria, Research Center Borstel, Leibniz Lung Center
Locations (2):
- Germany (2):
  - National and WHO-Supranational Reference Center for Mycobacteria, Research Center Borstel, Leibniz Lung Center, Borstel, Schleswig-Holstein
  - Klinik für Pneumologie, Universitätsklinikum Essen, Essen

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon reasonable request via contacting the prinicpal investigator.